CLINICAL TRIAL: NCT06737562
Title: Medico-economic Evaluation of Immediately Sequential Bilateral Cataract Surgery Compared With Delayed Sequential Cataract Surgery in France: a Multicenter Randomized Controlled Trial
Brief Title: Medico-economic Evaluation of Immediately Sequential Bilateral Cataract Surgery Compared With Delayed Sequential Cataract Surgery in France
Acronym: SIMCAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ASD_2023_5
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Cataract Bilateral; Bilateral Cataracts; Bilateral Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ISBCS (Experimental): Both eyes will be operated on during the same surgical procedure. Surgery will be performed in accordance with the iSBCS (International Society of Bilateral Cataract Surgeons) General Principles for Excellence in ISBCS (Immediate Sequential Bilateral Cataract Surgery) [12] by investigating ophthalmic surgeons or co-investigators with at least two years' experience in cataract surgery.
  Interventions: Procedure: Immediatly sequential bilateral cataract surgery
- DSBCS (Active Comparator): Only one eye will be operated on during the first surgiczal procedure. The second eye will be operated on during a second surgical procdure delayed from 3 weeks +/- 1 week. Surgeries will be performed according to current guidelines by investigating or co-investigating ophthalmic surgeons with at least two years' experience in cataract surgery.
  Interventions: Procedure: Delayed sequential bilateral cataract surgery

INTERVENTIONS:
Procedure: Immediatly sequential bilateral cataract surgery — Immediatly sequential bilateral cataract surgery
  Arms: ISBCS
Procedure: Delayed sequential bilateral cataract surgery — Delayed sequential bilateral cataract surgery : 3 weeks +/-1 week between the two procedures
  Arms: DSBCS

SUMMARY:
Cataracts are defined as opacification of all or part of the crystalline lens, resulting in reduced vision. It is a common disease in France, affecting more than one in five people over the age of 65, and almost two in three over the age of 85. Cataract treatment is exclusively surgical. In the case of bilateral cataracts, which account for 70% of cases, Delayed Sequential Bilateral Cataract Surgery (DSBCS), which involves operating on both eyes with an interval of a few weeks, is the reference treatment in France. The practice of DSBCS has long been justified by the need to reduce the risk of post-operative complications, essentially refractive error and bilateral endophthalmitis. Today, thanks to numerous technological advances in cataract surgery and new intraoperative standards, these complications have become exceptional. Since 2009, the International Society of Bilateral Cataract Surgeons (ISBCS) has issued a guide to best practice (the ''ISBCS General Principles for Excellence in ISBCS''), enabling surgery on both eyes to be performed on the same day in complete safety. As a result, Immediate Sequential Bilateral Cataract Surgery (ISBCS), which involves operating on both eyes on the same day, could be performed with no additional risk compared to SDBCS, while providing the same level of postoperative visual acuity. In view of these factors, we hypothesize that CCBIS would be an efficient alternative to DSBCS in cases of bilateral cataract, for the patient and his family, the hospital and the health insurance company. In addition, its adoption would reduce delays in access to treatment, thus promoting better access to care in the situation of growing demand for this treatment, particularly in areas with fewer medical facilities.

The aim of thisproject is to evaluate the associated costs and quality of life in comparison with CCBSD, based on a prospective, multicenter, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Indication for non-combined cataract surgery under local anaesthesia in both eyes
* Patient scheduled for outpatient cataract surgery
* Availability of a caregiver/accompanying person on the day of surgery and for the 1st day post-surgery
* Resident in France
* Speak and understand French
* Consent to participate in the study
* Affiliated or beneficiary of social security

Exclusion Criteria:

* Women of childbearing age
* Surgery scheduled under general anesthesia or combined with other eye surgeries
* Ocular tone > 24 mm Hg in at least one eye on day of inclusion
* Presence of risk factors for refractive error :

Presence of keratoconus confirmed by corneal topography Extreme axial eye length (< 21 mm or > 27 mm) High myopia with posterior staphyloma History of corneal surgery (LASIK, surface laser, radial keratotomy)

- Presence of risk factors for endophthalmitis : Ocular, periocular or adnexal infections Immunosuppression Uncontrolled diabetes

* Presence of risk factors for intraoperative complications Ocular, adnexal or anatomical abnormalities History of retinal detachment Lens dislocation or iridodonesis Black cataract or posterior polar cataract History of perforating or blunt ocular trauma
* Presence of risk factors for corneal edema (e.g. Fuchs' endothelial dystrophy)
* Presence of vision-related comorbidities (glaucoma, AMD, amblyopia, uveitis, etc.)
* Presence of diabetes with diabetic retinopathy or macular edema
* Patient unable to participate in follow-up (e.g., response to questionnaires)
* Presence of cognitive disorders that could affect the smooth running of surgery or response to questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Cost-utility of ISBCS compared to DSBCS | 3 months after index surgery (bilateral or on the first eye)
  Incremental cost-utility ratio calculated 3 months after the index surgery (1st surgery in the case of DSBCS), from the collective perspective.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Chu Morvan, Brest
  - Clinical Judge, Marseille
  - Cochin Hospital, Paris
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris